CLINICAL TRIAL: NCT06099795
Title: Evaluation of Concordance Between an Innovative Test on Exhaled Air (eBAM-CoV) and RT-PCR to Detect SARS-CoV-2 in Symptomatic Patients or Closed Contacts
Brief Title: Evaluation of Concordance Between Exhaled Air Test (eBAM-CoV) and RT-PCR to Detect SARS-CoV-2
Acronym: eBAM_CoV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: University of Nimes (Other); brains' laboratory sas, FRANCE (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IDIL/2022/VC-01
Record Dates: First submitted 2023-10-18; First posted 2023-10-25 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: SARS-CoV-2 Infection; COVID-19; Coronavirus
Keywords: Diagnostic Test Kits
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients likely to be affected by COVID-19 (Experimental): The study population consists of adult people who are likely to be affected by COVID-19 (symptomatic or close contacts) consulting for RT-PCR screening.
  Interventions: Device: eBAM Cov Testing

INTERVENTIONS:
Device: eBAM Cov Testing — Evaluation of presence/absence of infection with SARS-CoV-2 assessed by eBAM-CoV on air exhaled by the patient compared with the presence/absence of infection based on RT-PCR testing of nasopharyngeal swabs

SUMMARY:
During the COVID-19 pandemic, testing primarily relied on the use of nasopharyngeal swabs to detect the SARS-CoV-2 virus, responsible for the disease. However, this technique has several limitations, including the variable quality of swabs, its invasive nature, and arbitrariness in the choice of the number of cycles. Furthermore, it does not allow for the detection of viral proteins.

To overcome these limitations, researchers developed the eBAM-CoV test, patented for the detection of viral proteins in the exhaled air of COVID-19 patients. This portable device provides an immediate assessment of the "viral load" with both quantitative and qualitative results, showing promise for early virus detection.

The researchers hypothesize that the eBAM-CoV test is likely to exhibit a satisfactory concordance with the reference RT-PCR test in the detection of COVID-19, especially among symptomatic patients or closed contacts.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female patients over 18 years of age (≥)
* Suspected of being infected with COVID-19 (symptomatic or contact case) and consulting for RT-PCR screening.

Exclusion Criteria:

* Inability to understand the procedures to use the device
* Patient participating in an another interventional study
* Patient in exclusion period determined by another study
* Patient under court protection or guardianship
* Patient/trusted person/legal representative/family member for whom it is impossible to give informed information.
* Pregnant, parturient or breast-feeding patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Concordance between eBAM-Cov test and RT -PCR test to detect SARS-CoV -2 infection | Day 0
  Evaluate the performance of the eBAM-CoV test by measuring the concordance between the eBAM-CoV method and the reference RT-PCR method (known as the "gold standard") in detecting SARS-CoV-2 in subjects likely to be infected with COVID-19 (symptomatic or closed contacts).

SECONDARY OUTCOMES:
diagnostic performance of the eBAM-CoV test | Day 0
  Preliminarily assess the diagnostic performance of the eBAM-CoV test by measuring the sensitivity/specificity between the eBAM-CoV method and the reference RT-PCR method (known as the "gold standard") for detecting SARS-CoV-2 in subjects likely to be infected with COVID-19 (symptomatic or closed contact).
concentration of SARS-CoV-2 viral proteins | Day 0
  Correlation between the concentration of SARS-CoV-2 viral proteins assessed by the eBAM-CoV test (eBAM-Unit) and the mean number of copies of mRNA encoding a protein fraction of SARS-CoV-2 viral proteins assessed using the RT-PCR technique
Early detection of SARS-CoV-2 using eBAM-CoV test versus RT-PCR | Day 4
  Number of patients detected as positive by eBAM-CoV and negative by RT-PCR at Day 0 whose RT-PCR test becomes positive at Day 4
Concordance between eBAM-CoV test and antigenic test | Day 0
  Concordance between the eBAM-CoV method and the antigenic test in patients likely to be infected with COVID-19 and volunteering for a second nasopharyngeal swab

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Laboratoire Alphabio, Hôpital Européen Marseille, Marseille
  - CHU de NIMES, Nîmes

IPD SHARING:
Plan to Share IPD: No